CLINICAL TRIAL: NCT04926571
Title: Effect of Dexamethasone on Inpatient Mortality Among Hospitalized COVID-19 Patients
Brief Title: Dexamethasone and COVID-19 Inpatient Mortality
Status: Completed | Type: Observational
Sponsor: Aetion, Inc. (Other)
Responsible Party: Principal Investigator, Nicolle Gatto, Chief Science Officer, Aetion, Inc.
Other Study IDs: RQ004-1-20210610
Record Dates: First submitted 2021-06-11; First posted 2021-06-15 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Coronavirus
Keywords: treatment; dexamethasone; corticosteroid; mortality
MeSH Terms: conditions — Coronavirus Infections | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Dexamethasone versus non-users of corticosteroids
  Interventions: Drug: Dexamethasone Oral
- Dexamethasone versus non-users of dexamethasone
  Interventions: Drug: Dexamethasone Oral
- Dexamethasone versus methylprednisolone active comparator
  Interventions: Drug: Dexamethasone Oral

INTERVENTIONS:
Drug: Dexamethasone Oral — New users of Dexamethasone

SUMMARY:
The study aims to assess the effectiveness of dexamethasone initiation to reduce the risk of inpatient mortality within 28 days among US patients hospitalized with COVID-19 diagnosis or SARS-CoV-2 infection, overall and stratified by COVID-19 severity subgroups.

DETAILED DESCRIPTION:
This is a non-randomized, non-interventional study that is part of a research collaboration agreement between the US Food and Drug Administration (FDA) and Aetion to use real-world data to advance the understanding and the natural history of COVID-19 in specific patient populations, as well as treatment and diagnostic patterns during the coronavirus disease (COVID-19) pandemic.

This study compares inpatient mortality within 28 days among US patients hospitalized with COVID-19 diagnosis or SARS-CoV-2 infection who initiate dexamethasone treatment with a matched cohort of patients with 'standard of care' who are non-users of corticosteroids of interest (dexamethasone, prednisone, methylprednisolone, hydrocortisone). Patients are compared overall and and stratified by COVID-19 severity subgroups.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalized Patients with confirmed COVID-19 (diagnosis of U07.1 or positive or presumptive positive SARS-CoV-2 diagnostic laboratory test result) occurring between 21 days prior to the hospital admission date and the treatment index date.

Exclusion Criteria:

* No interaction with the healthcare system (medical encounter) in the 183 days prior to and including hospital admission (Day -183 to Day 0) to minimize the potential for misclassification of baseline covariates and/or new use
* No age or sex recorded in the 183 days prior to and including hospital admission (Day -183 to Day 0) as required for matching
* No geographic region recorded in 183 days prior to and including hospital admission (Day -183 to Day 0) as necessary to adjust for regional variation
* Any recorded use of any CSI (dispensing or remaining supply) in the 90-day washout prior to the treatment index date (Day T-90 to Day T-1) to satisfy new use definition
* Any record of a COVID-19 vaccine recorded on or any time prior to the treatment index date given that these patients are assumed to be selectively different (Day S to Day T)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized Patients with confirmed COVID-19 (diagnosis of U07.1 or positive or presumptive positive SARS-CoV-2 diagnostic laboratory test result) occurring between 21 days prior to the hospital admission date and the treatment index date.
  Patients will enter the cohort upon the admission date of the first qualifying inpatient hospitalization observed in the hospital chargemaster data. The first eligible cohort entry date is 01-April-2020, the date when the ICD-10 code for COVID-19 diagnosis was added.
Sampling Method: Probability Sample
Enrollment: 14105 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2021-08-27 (Actual); Study Completion 2021-08-27 (Actual)

PRIMARY OUTCOMES:
Mortality | 28 days
  Mortality within 28 days of admission

CONTACTS AND LOCATIONS:
Locations (1):
- Aetion, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Study results will report aggregated findings

DOCUMENTS (1):
  • Study Protocol (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/71/NCT04926571/Prot_000.pdf